CLINICAL TRIAL: NCT02131610
Title: Epigenetics Modifications and Subclinical Atherosclerosis in Obstructive Sleep Apnea: The EPIOSA Study
Brief Title: Epigenetics Modifications in Obstructive Sleep Apnea
Acronym: EPIOSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aragon Institute of Health Sciences (Other)
Collaborators: Instituto Aragones de Ciencias de la Salud (Other Government); Hospital Miguel Servet (Other)
Responsible Party: Sponsor
Other Study IDs: NCT01475421; PI12/02175 (Other: FISS)
Record Dates: First submitted 2014-04-16; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-04

CONDITIONS: Sleep Apnea; Snoring
Keywords: Sleep apnea; Obstructive sleep apnea; Subclinical atherosclerosis; Epigenetics; T cells
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — serum and plasma samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obstructive slep apnea patients: Patients with OSA
- Control group: Subjects without OSA

SUMMARY:
Changes in epigenetic regulation of genes involved in systemic inflammation and metabolic dysfunction in OSA are linked with accelerated cardiovascular morbidity.

DETAILED DESCRIPTION:
Design. EPIOSA is a 5-yr non-interventional longitudinal prospective study being conducted at the Sleep Clinic of the Hospital Miguel Servet, a large teaching hospital in Zaragoza (Spain). Following a baseline visit, subjects are to be followed-up at 3 months, and then every year.

Subject participation. The investigators will enroll a total 300 consecutive OSA male patients aged 20-60 yrs, with baseline apnea-hypopnea index ≥ 5 events per hour of sleep (AHI). In addition, 50 control subjects (AHI < 5) aged 20-60 yrs and matched by body mass index (BMI) are also to be recruited. Exclusion criteria will include any comorbid condition including alcohol and tobacco use.

Measurements: Routine clinical assessment, full sleep study, bilateral carotid ultrasonography, biochemistry, circulating inflammatory cytokines, T cell subsets and epigenetics studies at baseline and every year until at least 5 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 60

Exclusion Criteria:

* Any comorbid condition

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects that will be study because suspected OSA
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2013-03; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiovascular events according with or without the presence of epigenetics changes in pro-inflammatory genes | 5 years

SECONDARY OUTCOMES:
biomarkers in blood and urine that correlates with OSA severity which may serve also as markers of disease progression. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Marin, M.D., Principal Investigator — Hospital Miguel Servet
Locations (1):
- Hospital Miguel Servet, Zaragoza, Spain

REFERENCES:
- [Derived] Marin JM, Artal J, Martin T, Carrizo SJ, Andres M, Martin-Burriel I, Bolea R, Sanz A, Varona L, Godino J, Gallego B, Garcia-Erce JA, Villar I, Gil V, Forner M, Cubero JP, Ros L. Epigenetics modifications and Subclinical Atherosclerosis in Obstructive Sleep Apnea: The EPIOSA study. BMC Pulm Med. 2014 Jul 12;14:114. doi: 10.1186/1471-2466-14-114. PMID 25016368